CLINICAL TRIAL: NCT02567188
Title: A Study of MIRCERA in Participants With Chronic Kidney Disease Stage 3-4 and Not on Dialysis
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22439
Record Dates: First submitted 2015-09-28; First posted 2015-10-02 (Estimated); Results first posted 2015-12-30 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- Cohort of CKD Participants: Pre-dialysis participants with CKD treated with MIRCERA according to the current standard of care and in line with the current local summary of product characteristics were observed for maximum of 12 months.
  Interventions: Other: MIRCERA

INTERVENTIONS:
Other: MIRCERA

SUMMARY:
An observational, longitudinal, multi-center, non-interventional study in participants with chronic kidney disease (CKD) stage 3-4, assessed by Modification of Diet in Renal Disease (MDRD) to collect data regarding safety and efficacy in participants with pre-dialysis situation who are treated with MIRCERA in normal clinical environment.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants above 18 years of age
* Pre-dialysis participants with CKD stage 3-4 treated with MIRCERA and continue in the pre-dialysis state for the whole study period
* Estimated glomerular filteration rate (e-GFR) between 15-60 milliliter per minute (mL/min) (calculated)

Exclusion Criteria:

* Participants involved in interventional trials
* Participants with life expectancy less than 1 year
* Active malignancy
* Planned living kidney transplant within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with CKD Stage 3-4 treated with MIRCERA
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (18):
- Sweden (18):
  - Angeholm
  - Bollnäs
  - Eskilstuna
  - Gävle
  - Gothenburg
  - Huddinge
  - Jönköping
  - Karlshamn
  - Karlstad
  - Kristianstad
  - Linköping
  - Mölndal
  - Norrköping
  - Skövde
  - Stockholm
  - Umeå
  - Värnamo
  - Västervik

RESULTS

PARTICIPANT FLOW:
Groups:
- Chronic Kidney Disease (CKD) Participants: Pre-dialysis participants with CKD treated with MIRCERA according to the current standard of care and in line with the current local summary of product characteristics were observed for maximum of 12 months.
Period: Overall Study
Arm/Group | Chronic Kidney Disease (CKD) Participants
Started | 144
Completed | 109
Not Completed | 35
Not completed — Death | 10
Not completed — Terminated Mircera Treatment | 9
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Refused Treatment/ Did not Cooperate | 1
Not completed — Moved and Changed Clinic | 1
Not completed — Started Hemodialysis | 2
Not completed — Protocol Violation | 5

BASELINE CHARACTERISTICS:
Population: All enrolled participants with available data for baseline characteristics.
Groups:
- CKD Participants: Pre-dialysis participants with CKD treated with MIRCERA according to the current standard of care and in line with the current local summary of product characteristics were observed for maximum of 12 months.
Arm/Group | CKD Participants
Number analyzed (Participants) | 141
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.2 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64
  Male | 77

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reaching a Hemoglobin (Hb) Value of Greater Than (>) 100 and Less Than (<) 120 Grams Per Liter (gm/L) at Month 6 Before Inclusion
Time Frame: Pre-baseline (Month -6)
Population: All enrolled participants. Here, number of participants analyzed= participants with non-missing Hb assessment at specified time frame for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 125
percentage of participants | 56.8

2. Primary Outcome: Percentage of Participants Reaching a Hb Value of >100 and < 120 gm/L at Month 3 Before Inclusion
Time Frame: Pre-baseline (Month -3)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 116
percentage of participants | 56.0

3. Primary Outcome: Percentage of Participants Reaching a Hb Value of >100 and < 120 gm/L at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 139
percentage of participants | 42.4

4. Primary Outcome: Percentage of Participants Reaching a Hb Value of > 100 and < 120 gm/L at Month 3 After Inclusion
Time Frame: Month 3
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 122
percentage of participants | 41.0

5. Primary Outcome: Percentage of Participants Reaching a Hb Value of > 100 and < 120 gm/L at Month 6 After Inclusion
Time Frame: Month 6
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 113
percentage of participants | 41.6

6. Primary Outcome: Percentage of Participants Reaching a Hb Value of > 100 and < 120 gm/L at Month 9 After Inclusion
Time Frame: Month 9
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 106
percentage of participants | 33.0

7. Primary Outcome: Percentage of Participants Reaching a Hb Value of > 100 and < 120 gm/L at Month 12 After Inclusion
Time Frame: Month 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 110
percentage of participants | 45.5

8. Primary Outcome: Mean Hb Value at Month 6 Before Inclusion
Time Frame: Pre-baseline (Month -6)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 125
gm/L | 113.2 (11.7)

9. Secondary Outcome: Percentage of Participants With Change in MIRCERA Treatment
Description: Change in MIRCERA treatment included changes in dose, frequency, and route of administration.
Time Frame: Months 3, 6, 9, and 12
Population: All enrolled participants. Here, number of participants analyzed= participants evaluable for this outcome measure. n = number of participants evaluable at the specified time frame.
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 130
percentage of participants
  Month 3 (n= 130) | 43.1
  Month 6 (n= 117): number analyzed (Participants) | 117
  Month 6 (n= 117) | 30.8
  Month 9 (n= 110): number analyzed (Participants) | 110
  Month 9 (n= 110) | 22.7
  Month 12 (n= 112): number analyzed (Participants) | 112
  Month 12 (n= 112) | 23.2

10. Secondary Outcome: Percentage of Participants With Number of MIRCERA Dose Changes
Time Frame: Baseline to Month 12
Population: All enrolled participants. Here, number of participants analyzed= participants with available data for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 91
percentage of participants
  No change | 26.4
  One change | 41.8
  Two changes | 17.6
  Three changes | 13.2
  Four changes | 1.1

11. Secondary Outcome: Correlation of Hb Levels With Underlying Disease
Time Frame: Baseline to 12 months
Population: The units usage at and between study centres did change during the study and therefore no descriptive statistics could be performed on the laboratory variables.
Arm/Group | CKD Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Correlation of Hb Levels With Levels of Inflammation
Time Frame: Baseline to 12 months
Population: as for outcome 11
Arm/Group | CKD Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Percentage of Participants With Changes in Iron Supplement
Description: Percentage of participants who had any change in their iron supplement medication at a specified visit were reported.
Time Frame: Pre-baseline (Months -6 and -3), baseline, Months 3, 6, 9 and 12
Population: All enrolled participants. Here, number of participants analyzed= participants evaluable for this outcome measure and n= participants evaluable for specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | Cohort of CKD Participants
Number analyzed (Participants) | 142
percentage of participants
  Pre-baseline (Month -6) (n= 134): number analyzed (Participants) | 134
  Pre-baseline (Month -6) (n= 134) | 31.3
  Pre-baseline (Month -3) (n= 125): number analyzed (Participants) | 125
  Pre-baseline (Month -3) (n= 125) | 12.8
  Baseline (n= 142) | 15.5
  Month 3 (n= 130): number analyzed (Participants) | 130
  Month 3 (n= 130) | 11.5
  Month 6 (n= 115): number analyzed (Participants) | 115
  Month 6 (n= 115) | 13.0
  Month 9 (n= 109): number analyzed (Participants) | 109
  Month 9 (n= 109) | 9.2
  Month 12 (n= 112): number analyzed (Participants) | 112
  Month 12 (n= 112) | 12.5

14. Primary Outcome: Mean Hb Value at Month 3 Before Inclusion
Time Frame: Pre-baseline (Month -3)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 116
gm/L | 112.6 (13.2)

15. Primary Outcome: Mean Hb Value at Baseline
Time Frame: Baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 139
gm/L | 117.5 (15.0)

16. Primary Outcome: Mean Hb Value at Month 3 After Inclusion
Time Frame: Month 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 122
gm/L | 120.2 (13.2)

17. Primary Outcome: Mean Hb Value at Month 6 After Inclusion
Time Frame: Month 6
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 113
gm/L | 120.0 (13.8)

18. Primary Outcome: Mean Hb Value at Month 9 After Inclusion
Time Frame: Month 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 106
gm/L | 120.0 (14.3)

19. Primary Outcome: Mean Hb Value at Month 12 After Inclusion
Time Frame: Month 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: gm/L
Arm/Group | CKD Participants
Number analyzed (Participants) | 110
gm/L | 118.4 (12.8)

20. Primary Outcome: Percentage of Participants With Hb Fluctuation From Pre-Baseline (Month -6) to Baseline
Description: Hb fluctuation was defined as change in Hb value >15 gm/L between 2 visits.
Time Frame: Pre-baseline (Month -6) to Baseline
Population: All enrolled participants. Here, number of participants analyzed= participants with at least 2 non-missing Hb assessments between pre-baseline (Month -6) and baseline.
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 126
percentage of participants | 36.5

21. Primary Outcome: Percentage of Participants With Hb Fluctuation From Baseline to Month 12
Description: Hb fluctuation was defined as change in Hb value >15 gm/L between 2 visits.
Time Frame: Baseline to Month 12
Population: All enrolled participants. Here, number of participants analyzed= participants with at least 2 non-missing Hb assessments between baseline and Month 12.
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 117
percentage of participants | 43.6

22. Secondary Outcome: Percentage of Participants With Changes in Immunosuppressive Treatment
Description: Percentage of participants who had any change in their immunosuppressive medication at a specified visit were reported.
Time Frame: Pre-baseline (Months -6 and -3), baseline, Months 3, 6, 9 and 12
Population: All enrolled participants. Here, number of participants analyzed = participants evaluable for this outcome measure and n= participants evaluable for specified time points.
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 142
percentage of participants
  Pre-baseline (Month -6) (n= 135): number analyzed (Participants) | 135
  Pre-baseline (Month -6) (n= 135) | 23.0
  Pre-baseline (Month -3) (n= 125): number analyzed (Participants) | 125
  Pre-baseline (Month -3) (n= 125) | 4.0
  Baseline (n= 142) | 5.6
  Month 3 (n= 129): number analyzed (Participants) | 129
  Month 3 (n= 129) | 8.5
  Month 6 (n= 114): number analyzed (Participants) | 114
  Month 6 (n= 114) | 8.8
  Month 9 (n= 109): number analyzed (Participants) | 109
  Month 9 (n= 109) | 2.8
  Month 12 (n= 111): number analyzed (Participants) | 111
  Month 12 (n= 111) | 5.4

23. Secondary Outcome: Percentage of Participants With Changes in Antihypertensive Treatment
Description: Percentage of participants who had any change in their antihypertensive medication at a specified visit were reported.
Time Frame: Pre-baseline (Months -6 and -3), baseline, Months 3, 6, 9 and 12
Population: as for outcome 22
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 141
percentage of participants
  Pre-baseline (Month -6) (n= 135): number analyzed (Participants) | 135
  Pre-baseline (Month -6) (n= 135) | 78.5
  Pre-baseline (Month -3) (n= 125): number analyzed (Participants) | 125
  Pre-baseline (Month -3) (n= 125) | 22.4
  Baseline (n= 141) | 22.7
  Month 3 (n= 130): number analyzed (Participants) | 130
  Month 3 (n= 130) | 12.3
  Month 6 (n= 115): number analyzed (Participants) | 115
  Month 6 (n= 115) | 13.0
  Month 9 (n= 109): number analyzed (Participants) | 109
  Month 9 (n= 109) | 16.5
  Month 12 (n= 111): number analyzed (Participants) | 111
  Month 12 (n= 111) | 19.8

24. Secondary Outcome: Number of Participants With Different Medication Treatment
Description: Number of participants who were receiving different treatments (antihypertensive, immunosuppressive, iron supplements, and others) before and/or after baseline were reported. Same participant could be reported in more than one category.
Time Frame: Pre-baseline (Month -6) to Month 12
Population: All enrolled participants. Here, number of participants analyzed= participants evaluable for this outcome measure.
Measure: Number; unit: participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 142
participants
  Anti-hypertensive treatment | 123
  Immunosuppressive treatment | 35
  Iron treatment | 71
  Other treatment | 55

25. Secondary Outcome: Percentage of Participants Who Required Blood Transfusion
Time Frame: Pre-baseline (Months -6 and -3), baseline, Months 3, 6, 9 and 12
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 142
percentage of participants
  Pre-baseline (Month -6) (n= 136): number analyzed (Participants) | 136
  Pre-baseline (Month -6) (n= 136) | 0
  Pre-baseline (Month -3) (n= 128): number analyzed (Participants) | 128
  Pre-baseline (Month -3) (n= 128) | 2.3
  Baseline (n= 142) | 5.6
  Month 3 (n= 131): number analyzed (Participants) | 131
  Month 3 (n= 131) | 1.5
  Month 6 (n= 115): number analyzed (Participants) | 115
  Month 6 (n= 115) | 1.7
  Month 9 (n= 109): number analyzed (Participants) | 109
  Month 9 (n= 109) | 3.7
  Month 12 (n= 110): number analyzed (Participants) | 110
  Month 12 (n= 110) | 1.8

26. Secondary Outcome: Percentage of Participants Who Required Renal Replacement Therapy
Description: Renal replacement therapy was defined as hemodialysis and peritoneal dialysis.
Time Frame: Months 3, 6, 9, and 12
Population: as for outcome 13
Measure: Number; unit: percentage of participants
Arm/Group | CKD Participants
Number analyzed (Participants) | 130
percentage of participants
  Hemodialysis done: Month 3 (n= 130) | 0.8
  Hemodialysis done: Month 6 (n= 113): number analyzed (Participants) | 113
  Hemodialysis done: Month 6 (n= 113) | 0.9
  Hemodialysis done: Month 9 (n= 107): number analyzed (Participants) | 107
  Hemodialysis done: Month 9 (n= 107) | 0.9
  Hemodialysis done: Month 12 (n= 110): number analyzed (Participants) | 110
  Hemodialysis done: Month 12 (n= 110) | 1.8
  Peritoneal dialysis done: Month 3 (n= 130) | 0.8
  Peritoneal dialysis done: Month 6 (n= 113): number analyzed (Participants) | 113
  Peritoneal dialysis done: Month 6 (n= 113) | 0
  Peritoneal dialysis done: Month 9 (n= 107): number analyzed (Participants) | 107
  Peritoneal dialysis done: Month 9 (n= 107) | 0.9
  Peritoneal dialysis done: Month 12 (n= 110): number analyzed (Participants) | 110
  Peritoneal dialysis done: Month 12 (n= 110) | 1.8

ADVERSE EVENTS:
Time Frame: Pre-baseline (Month -6) to Month 12
Description: All enrolled participants with data recorded for adverse events were included.
Arm/Group | CKD Participants
Serious Adverse Events (participants affected / at risk) | 0/141
Other Adverse Events (participants affected / at risk) | 1/141
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CKD Participants (N=141)
Skin Reaction (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but only after the first publication or presentation that involves the Overall Study. The sponsor may request that the confidential information be deleted and/or the publication to be postponed inorder to present the Sponsor's intellectual property rights.